CLINICAL TRIAL: NCT02600234
Title: REDUCE LAP-HF RANDOMIZED TRIAL I: A Study to Evaluate the Corvia Medical, Inc. IASD® System II to REDUCE Elevated Left Atrial Pressure in Patients With Heart Failure
Brief Title: REDUCE LAP-HF RANDOMIZED TRIAL I
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corvia Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1501
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment with Inter-Atrial Shunt Device (Experimental): Once all study criteria have been met, if randomized to this arm, patients will receive the IASD implant.
  Interventions: Device: Inter-Atrial Shunt Device
- Control (Placebo Comparator): Once all study criteria have been met, if randomized to this arm, patients will not receive the implant. They will undergo an intracardiac echo only, with the option to crossover at 1 year.
  Interventions: Other: Intracardiac Echo

INTERVENTIONS:
Device: Inter-Atrial Shunt Device — An implantable device placed in the interatrial septum
  Other Names: IASD
  Arms: Treatment with Inter-Atrial Shunt Device
Other: Intracardiac Echo — Patients randomized to the control arm will undergo intra cardiac echocardiography, with examination of the atrial septum and left atrial appendage.
  Arms: Control

SUMMARY:
A study to evaluate the Corvia Medical, Inc. IASD® System II to REDUCE Elevated Left Atrial Pressure in Patients with Heart Failure.

DETAILED DESCRIPTION:
The primary objective of this randomized controlled clinical study is to evaluate the peri-procedural safety and potential effectiveness (mechanistic effect) of implanting the IASD System II in heart failure patients with an LV ejection fraction >40%, elevated left sided filling pressures, and who remain symptomatic despite optimal Guideline Directed Medical Therapy (GDMT). Clinical outcomes will also be evaluated.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic symptomatic Heart Failure
* Ongoing stable GDMT HF management and management of potential comorbidities
* Age ≥ 40 years old
* LV ejection fraction ≥ 40% within the past 3 months, without previously documented ejection fraction <30%.
* Elevated left atrial pressure with a gradient compared to right atrial pressure (RAP) documented by end-expiratory PCWP during supine ergometer exercise ≥ 25mm Hg, and greater than RAP by ≥ 5 mm Hg

Key Exclusion Criteria:

* MI and/or percutaneous cardiac intervention within past 3 months; CABG in past 3 months, or current indication for coronary revascularization
* Cardiac Resynchronization Therapy initiated within the past 6 months
* Severe heart failure
* Inability to perform 6 minute walk test (distance < 50 m), OR 6 minute walk test > 600m
* History of stroke, transient ischemic attack (TIA), deep vein thrombosis (DVT), or pulmonary emboli within the past 6 months
* Presence of significant valve disease
* Known clinically significant untreated carotid artery stenosis
* Currently requiring dialysis; or estimated-GFR <25ml/min/1.73 m2 by CKD-Epi equation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Peri-procedural, and 1 month Major Adverse Cardiac, Cerebrovascular, and Renal Events (MACCRE) | 1 Month Post Implant
  The primary safety outcome measure is the incidence of one or more of the following major adverse cardiac, cerebrovascular embolic, or renal events (MACCRE) defined as:
  1. Cardiovascular death through 1-month post implant;
  2. Embolic stroke through 1-months post implant;
  3. Device and or procedure related adverse cardiac events through 1-month post implant;
  4. New onset or worsening of kidney dysfunction (defined as eGFR decrease of > 20 ml/min) through 1-month post implant
Change in supine exercise pulmonary capillary wedge pressure (PCWP) | 1 Month Post Implant
  Change in supine exercise pulmonary capillary wedge pressure (PCWP), as assessed by an independent blinded hemodynamic core laboratory, across the four values measured at each visit (values at 20W, 40W, 60W and 80W).

SECONDARY OUTCOMES:
Change in exercise PEAK pulmonary capillary wedge pressure (PCWP) from baseline | 1 Month
Cardiovascular death | 12 Months
Rate of total (first plus recurrent) HF admissions/emergency clinic visits or acute care facilities for IV diuresis for HF | 12 Months
Change in Quality Of Life Questionnaire (EQ-5D) | 12 Months
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ score) | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Shah, MD, Principal Investigator — Northwestern University
Locations (21):
- United States (17):
  - University of Arizona College of Medicine, Tucson, Arizona
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - Evanston Northshore Healthcare, Evanston, Illinois
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center/NewYork Presbyterian Hospital, New York, New York
  - Mt. Sinai Hospital, New York, New York
  - New York University, New York, New York
  - Wake Forest, Winston-Salem, North Carolina
  - Ohio Health, Columbus, Ohio
  - Ohio State University College of Medicine, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
- The Alfred Hospital, Melbourne, Australia
- OLVZ Aalst, Aalst, Belgium
- UMC Groningen, Groningen, Netherlands
- Golden Jubilee Hospital, Glasgow, United Kingdom

REFERENCES:
- [Derived] Litwin SE, Komtebedde J, Borlaug BA, Kaye DM, Hasenfubeta G, Kawash R, Hoendermis E, Hummel SL, Cikes M, Gustafsson F, Chung ES, Mohan RC, Sverdlov AL, Swarup V, Winkler S, Hayward CS, Bergmann MW, Bugger H, McKenzie S, Nair A, Rieth A, Burkhoff D, Cutlip DE, Solomon SD, van Veldhuisen DJ, Leon MB, Shah SJ. Long term safety and outcomes after atrial shunting for heart failure with preserved or mildly reduced ejection fraction: 5-year and 3-year follow-up in the REDUCE LAP-HF I and II trials. Am Heart J. 2024 Dec;278:106-116. doi: 10.1016/j.ahj.2024.08.014. Epub 2024 Sep 3. PMID 39237070
- [Derived] Obokata M, Reddy YNV, Shah SJ, Kaye DM, Gustafsson F, Hasenfubeta G, Hoendermis E, Litwin SE, Komtebedde J, Lam C, Burkhoff D, Borlaug BA. Effects of Interatrial Shunt on Pulmonary Vascular Function in Heart Failure With Preserved Ejection Fraction. J Am Coll Cardiol. 2019 Nov 26;74(21):2539-2550. doi: 10.1016/j.jacc.2019.08.1062. PMID 31753198
- [Derived] Shah SJ, Feldman T, Ricciardi MJ, Kahwash R, Lilly S, Litwin S, Nielsen CD, van der Harst P, Hoendermis E, Penicka M, Bartunek J, Fail PS, Kaye DM, Walton A, Petrie MC, Walker N, Basuray A, Yakubov S, Hummel SL, Chetcuti S, Forde-McLean R, Herrmann HC, Burkhoff D, Massaro JM, Cleland JGF, Mauri L. One-Year Safety and Clinical Outcomes of a Transcatheter Interatrial Shunt Device for the Treatment of Heart Failure With Preserved Ejection Fraction in the Reduce Elevated Left Atrial Pressure in Patients With Heart Failure (REDUCE LAP-HF I) Trial: A Randomized Clinical Trial. JAMA Cardiol. 2018 Oct 1;3(10):968-977. doi: 10.1001/jamacardio.2018.2936. PMID 30167646
- [Derived] Feldman T, Mauri L, Kahwash R, Litwin S, Ricciardi MJ, van der Harst P, Penicka M, Fail PS, Kaye DM, Petrie MC, Basuray A, Hummel SL, Forde-McLean R, Nielsen CD, Lilly S, Massaro JM, Burkhoff D, Shah SJ; REDUCE LAP-HF I Investigators and Study Coordinators. Transcatheter Interatrial Shunt Device for the Treatment of Heart Failure With Preserved Ejection Fraction (REDUCE LAP-HF I [Reduce Elevated Left Atrial Pressure in Patients With Heart Failure]): A Phase 2, Randomized, Sham-Controlled Trial. Circulation. 2018 Jan 23;137(4):364-375. doi: 10.1161/CIRCULATIONAHA.117.032094. Epub 2017 Nov 15. PMID 29142012
- [Derived] Feldman T, Komtebedde J, Burkhoff D, Massaro J, Maurer MS, Leon MB, Kaye D, Silvestry FE, Cleland JG, Kitzman D, Kubo SH, Van Veldhuisen DJ, Kleber F, Trochu JN, Auricchio A, Gustafsson F, Hasenfubeta G, Ponikowski P, Filippatos G, Mauri L, Shah SJ. Transcatheter Interatrial Shunt Device for the Treatment of Heart Failure: Rationale and Design of the Randomized Trial to REDUCE Elevated Left Atrial Pressure in Heart Failure (REDUCE LAP-HF I). Circ Heart Fail. 2016 Jul;9(7):e003025. doi: 10.1161/CIRCHEARTFAILURE.116.003025. PMID 27330010